CLINICAL TRIAL: NCT01328691
Title: Prognostic Factors for Korean Patients With Renal Cell Carcinoma and Venous Tumor Thrombus Extension: Application of the New 2009 TNM Staging System
Brief Title: Prognostic Factor for Renal Cell Carcinoma (RCC) With Venous Tumor Thrombus
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Cheol Kwak / M.D., Ph.D., Seoul National University Hospital
Other Study IDs: MCCho5
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Carcinoma, Renal Cell; Thrombus
Keywords: Carcinoma, Renal Cell; thrombus; body mass index; grade
MeSH Terms: conditions — Carcinoma, Renal Cell; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Renal cell carcinoma (RCC) has its propensity to invade the venous system, with extension into the renal vein and the inferior vena cava (IVC) in 23% and 7%, respectively. Despite advances in radiation, chemotherapy, and immunotherapy the reference standard for RCC with tumor thrombus remains surgical resection. However, the 5-year survival rate for patients who have RCC with venous tumor thrombus treated with radical nephrectomy and tumor thrombectomy is only 35% - 45%, despite the developments in surgical technique and perioperative care. Furthermore, even the 5-year survival rate for the patients without the evidence of nodal or distant metastasis at presentation is just 45% - 65%.

The outcome prediction for RCC remains controversial, and although many parameters have been tested for prognostic significance, only a few have achieved widespread acceptance in clinical practice. Currently, pathologic stage (T stage), lymph node status (N stage) and histologic grade represent the main prognostic variables in the patients with RCC and venous tumor thrombus. Accordingly, the American Joint Committee on Cancer (AJCC) TNM classification is regularly revised and, recently, a new 2009 AJCC TNM stage classification system has been proposed.

RCC is more prevalent in developed countries, such as Europe and North America. It is relatively less common in Asia; however, the incidence in these regions appears to have risen over the past decade. Recently, a few series have suggested that racial or ethnic differences in survival persist after controlling for age and stage in some cancers. In the case of renal cell carcinoma, it has been demonstrated that the malignancy diagnosed in various ethnic groups had different clinical characteristics: the presenting symptoms, the course of disease, and the outcome after standard treatment varied significantly between patients of Caucasian, Hispanic, African-American, and Asian backgrounds. A recent study has reported that race as well as established factors has an impact on survival in patients with RCC and Asian Pacific Islander ethnicity was predictive of improved overall or cancer specific survival.

Up to date, there was sparse data on surgical outcome and prognostic factors of survival after radical nephrectomy and thrombectomy in an Asian population with RCC and venous tumor thrombus, while most studies have been performed in Western countries. The aim of the present study was to address the surgical outcome after radical nephrectomy with thrombectomy and to evaluate the prognostic factors influencing on survival in Korean patients with RCC and tumor thrombus extension into renal vein or IVC, labeled as T3a and T3b-c by the newly revised 2009 AJCC TNM staging system, respectively.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* patients with RCC and venous tumor thrombus who underwent radical nephrectomy and thrombectomy

Exclusion Criteria:

* von Hippel-Lindau disease
* tuberous sclerosis syndrome
* Wilms' tumor
* synchronous bilateral tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From Feburary 1988 to April 2009, a total of 118 patients with RCC and venous tumor thrombus who underwent radical nephrectomy and thrombectomy at our tertiary referal center
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cancer-specific survival | Five years

SECONDARY OUTCOMES:
Recurrence-free survival | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Kwak, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea